CLINICAL TRIAL: NCT04639492
Title: Evaluating the Effect and Safety of Postbiotic MBS and Metformin Combination on Gut Microbiota and Symptom in Patients With Diabetes
Brief Title: Postbiotic MBS and Metformin Combination in Patients With T2DM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Microbio Co Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MBSCLAS01
Record Dates: First submitted 2020-11-10; First posted 2020-11-20 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2023-01

CONDITIONS: Type-II Diabetes
Keywords: Diabetes Mellitus (DM); diabetes; T2DM; MBS; microbial
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MBS oral solution (Experimental): fermented soybean extract-MBS
  Interventions: Dietary Supplement: MBS oral solution

INTERVENTIONS:
Dietary Supplement: MBS oral solution — Oral BIDAC, twice a day before breakfast and dinner times

SUMMARY:
The primary objective is to evaluate the effect of MBS treatment in human subjects, and to validate its impact on intestinal flora and diabetes symptoms on diabetic patients undertaking metformin. The scientific data collected will be referenced for future product development.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subject who aged from 20 to 70.
2. BMI in between 18.5 and 35 kg/m2 inclusively.
3. Fasting blood sugar ≥ 126 mg/dL, and confirmed diagnosis of type-II diabetes.
4. 30 days prior to the screening visit (V1), HbA1c is steadily maintained in between 7-10% by medication.
5. Prior to the screening visit (V1), subjects have been regularly taken 500-200 mg/day for at least 90 days.

Exclusion Criteria:

1. Pregnant or breastfeeding women or female subjects plan to enter pregnancy during study period.
2. Subjects who are allergic to soy or products containing it.
3. At investigator's discretion, subjects are unlikely to comply with study procedures due to a history of alcohol or drug addiction.
4. Subjects on vegetarian diet or other special diets (eg. Ketogenic or gluten-free diets).
5. Subjects have ongoing participation in another clinical trial that involves the use of investigational drugs, medical devices, dietary supplements, and/or cosmetics.
6. Subject with impaired renal function confirmed by Serum Total Bilirubin ≥ 1.5 upper limit of normal [ULN], Aspartate Transaminase/ Alanine Transaminase (AST/ALT) ≥ 2 ULN, Creatinine ≥ 2 ULN or eGFR <60 mL/min/1.73 m^2.
7. Subjects who have been diagnosed with malignant tumors within five (5) years before the screening visit (V1) with exception to subjects with topical cancer but show significant recovery following investigator's assessment, such as basal or squamous cell skin cancer, superficial bladder cancer, or prostate or cervix or carcinoma in situ of the breast.
8. 30 days prior to screening visit (V1), subjects have taken antibiotics, synthetic drugs (Sulfonamides, Fluoroquinolone, etc.), anti-fungal or anti-viral medication but not limited to topical forms for use in skin application.
9. Within 14 days prior to screening visit (V1), subjects have taken products or supplements that contain probiotics or prebiotics.
10. Within 14 days prior to screening visit (V1), subjects experience diarrhea caused by gastrointestinal infection (3 times of watery stool within 24 hours).
11. Within14 days prior to screening visit (V1), subjects have taken steroids, immunosuppressant, and/or inflammatory medicines.
12. Subjects took or intend to take medications other than metformin that may affect intestinal flora within 30 days prior to screening visit, during screening period or whole trial period. Examples of this kind of medication include DPP-4 inhibitors, GLP-1 receptor agonists, acarbose, hypoglycemic sulfonamides, thiazolidinediones, SGLT2 inhibitors, and insulin.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-09-23 (Actual)

PRIMARY OUTCOMES:
Post-treatment changes of intestinal flora | 4, 8,12 weeks post-treatment
  Post-treatment changes from baseline in microbial composition, abundance, variation of subject's intestinal flora at 4, 8, 12 weeks.

SECONDARY OUTCOMES:
Post-treatment changes from baseline in fasting plasma glucose at 12 weeks | 12 weeks post-treatment
Post-treatment changes from baseline in HbA1c at 12 weeks | 12 weeks post-treatment
Post-treatment changes from baseline in HOMA-IR at 12 weeks | 12 weeks post-treatment
Post-treatment changes from baseline in blood lipids composition at 12 weeks | 12 weeks post-treatment
  Changes of triglyceride, high-density lipoprotein (HDL), and low-density lipoprotein (LDL)
Post-treatment changes from baseline in immune factors at 12 weeks | 12 weeks post-treatment
  Changes of CRP, IL6, TNF-α expression
Incidence of treatment-emergent adverse events(TEAE) | 12 weeks post-treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Microbio Investigative Site, Taipei, Taiwan